CLINICAL TRIAL: NCT02162875
Title: Parasitologic Impact of Different Mass Drug Administration Strategies Against Schistosoma Mansoni in Endemic Areas of Mwanza Region, Tanzania, Where Prevalence is 25% or Above
Brief Title: Schistosoma Mansoni in Mwanza Region, Tanzania
Acronym: SCORE_PAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Responsible Party: Principal Investigator, Pascal Magnussen, Associate Professor, DBL -Institute for Health Research and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAN-score; BMGF (Other Grant/Funding Number: BMGF)
Record Dates: First submitted 2014-05-26; First posted 2014-06-13 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Schistosoma Mansoni
Keywords: Schistosoma mansoni; treatment; school children; adults
MeSH Terms: conditions — Schistosomiasis | interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- MDA once a year (Experimental): Community wide treatment (CWT) once a year for four years with single dose praziquantel 40mg/kg
  Interventions: Drug: Praziquantel
- MDA 2nd year CWT follwed by 2 years SBT (Experimental): Treatment with praziquantel as arm 1 given by two years of community wide treatment (CWT) followed by two years of school-based treatment (SBT)
  Interventions: Drug: Praziquantel
- Praziquantel every second year CWT (Experimental): Treatment with praziquantel given every second year as CWT
  Interventions: Drug: Praziquantel
- MDA once a year SBT (Experimental): Treatment with praziquantel as above given as 4 years of SBT
  Interventions: Drug: Praziquantel
- MDA given for 2 years as SBT (Experimental): Treatment with praziquantel as above given for 2 years as SBT followed by 2 years without MDA
  Interventions: Drug: Praziquantel
- MDA as SBT 1year and 1 year without MDA (Experimental): Treatment with praziquantel given as one years of SBT alternating with one year without treatment
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Praziquantel — Six different treatment strategies with praziquantel
  Other Names: no other drugs

SUMMARY:
The objective of this study is to determine the strategy for mass drug administration (MDA) which provides the greatest reductions in prevalence and intensity of Schistosoma mansoni in school-aged children after 4 years of intervention.

DETAILED DESCRIPTION:
Intestinal schistosomiasis is caused by the blood-dwelling flatworm Schistosoma mansoni. Despite the increasing focus on the use of praziquantel against schistosomiasis infections for the last three decades many areas in Sub-Saharan Africa still have high prevalences and intensities of schistosomiasis especially among school-age children. This is true for the area of Mwanza Region of Tanzania adjacent to Lake Victoria. The study is a six arm study and includes 150 communities (25 in each arm). From each community 100 school children (aged 9-12 years), 100 first year students (aged 7-8 years) and 50 adults (aged 20-55 years) are included, diagnosed and treated with praziquantel using strategies composing of a mixture of community wide treatment (CWT), school-based treatment (SBT) and years without treatment (-T). The 100 school children provided stool specimens on three consecutive days, while the 100 first year students and 50 adults with few exceptions only provided one specimen. The treatment strategies during the 4 years for the different arms are as follows: Arm 1: CWT, CWT, CWT, CWT; Arm 2: CWT, CWT, SBT, SBT; Arm 3: CWT, CWT -T, -T; Arm 4: SBT, SBT, SBT, SBT; Arm 5: SBT, SBT, -T, -T; Arm 6: SBT, -T, SBT, -T.

ELIGIBILITY:
Inclusion Criteria:

-All school children and adults who consent to participate can be included

Exclusion Criteria:

-Those not consenting or with any chronic disease not related to schistosomiasis will be excluded

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37500 (Estimated)
Dates: Start 2011-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Effect of Mass drug administration on prevalence and intensity of Schistosoma mansoni among children and adults | May -October 2016 (5 months)
  Prevalence and intensity of Schistosoma mansoni

SECONDARY OUTCOMES:
Mass drug administration coverage | May -October 2016 (5 months)
  Coverage of treatment

OTHER OUTCOMES:
Cost of different treatment arm | May-October 2016 (5 months)
  Cost of different treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Safari Kinung'hi, PhD, Principal Investigator — National Institute for Medical Research, Mwanza Research Centre
Locations (1):
- National Institute for Mediacal Research, Mwanza, Kagera, Tanzania

IPD SHARING:
Plan to Share IPD: No